CLINICAL TRIAL: NCT04431388
Title: Analgesic Effectiveness of the Serratus-intercostal Plane Block Versus Quadratus Lumborum Block in Nephrectomy: Randomized Study
Brief Title: Serratus-intercostal Plane Block Versus Quadratus Lumborum Block in Nephrectomy: Randomized Study
Status: Completed | Type: Observational
Sponsor: Hospital Medina del Campo (Other)
Responsible Party: Principal Investigator, María Teresa Fernandez, Principal Investigator, Hospital Medina del Campo
Other Study IDs: CASVE-NM-20-434; 2020-000779-19 (EudraCT Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Kidney Injury
Keywords: postoperative analgesia; fascial blocks; nephectomy
MeSH Terms: interventions — Ultrasonography; Equipment and Supplies; Levobupivacaine; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- SIPB (block): Patients undergone nephectomy and who received SIPB as analgesia
  Interventions: Device: ultrasound device; Drug: Levobupivacaine
- QL block: Patients undergone nephectomy and who received QL as analgesia
  Interventions: Device: ultrasound device; Drug: Levobupivacaine
- control: Patients undergone nephrectomy who didn´t receive regional anesthesia

INTERVENTIONS:
Device: ultrasound device — We performe a differnt analgesic techniques to know if some of then are better
  Other Names: device
  Groups: QL block; SIPB (block)
Drug: Levobupivacaine — using the same AL
  Other Names: drug
  Groups: QL block; SIPB (block)

SUMMARY:
Performing the nephrectomy by laparoscopy has decrease the incidence of postoperative pain, but there are still some patients who describe a severe pain after this surgery. Regional techniques allow a better recovery quality and adequate- managed pain control.

DETAILED DESCRIPTION:
Adequate control of pain in patients with nephrectomy is a challenge for the anesthesiologist who must achieve an early recovery with minimal adverse effects. Within a multimodal strategy, the work hypothesis is based on comparing the analgesic efficacy of two regional techniques in patients undergoing nephrectomy, in terms of quality of postoperative recovery, pain control, absence of adverse effects and ease of performance.

ELIGIBILITY:
Inclusion Criteria:

* signature of informed consent
* age > 18 years
* ASA risk scale < IV
* Scheduled to nephrectomy.

Exclusion Criteria:

* Patients with cognitive impairment or inability to sign informed consent,
* Refused to participate
* Hypersensitivity to the drugs used
* contraindication of regional technique (coagulopathy, infection)
* history of chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 80 patients (40 in each group) has been calculated assuming that we intend to confirm a 15% improvement in pain control and postoperative recovery in the serratus-intercostal plane block group.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
pain control and quality life.Numeric rating scale (NRS) | "24 postoperative hours"
  To assess whether SIPB is superior in pain control
QoR15 | "24hours"
  Postoperative quality recovery

SECONDARY OUTCOMES:
Opioids consumption | "48 hours"
  Second outcomes was to know the consumption of intaoperative fentanyl and postoperative morphine and their side effects
Side effects | "24hours"
  We assessed the side effects of opioids

OTHER OUTCOMES:
control | "24 hours"
  Third outcome will be to know if both blocks control pain better than control group

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Fernandez, Study Chair — Hospital Medina del Campo
Locations (1):
- María Teresa Fernandez, Valladolid, VA, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corso RM, Piraccini E, Sorbello M, Bellantonio D, Tedesco M. Ultrasound-guided transmuscular quadratus lumborum block for perioperative analgesia in open nephrectomy. Minerva Anestesiol. 2017 Dec;83(12):1334-1335. doi: 10.23736/S0375-9393.17.12167-X. Epub 2017 Jul 5. No abstract available. PMID 28679202
- [Background] Corso RM, Piraccini E, Sorbello M, Bellantonio D, Tedesco M. Transmuscular quadratus lumborum block versus serratus-intercostal interfascial plane block: the game has just begun. Minerva Anestesiol. 2018 Jul;84(7):873-874. doi: 10.23736/S0375-9393.18.12849-5. Epub 2018 Mar 27. No abstract available. PMID 29589427
- [Background] Fernandez Martin MT, Lopez Alvarez S, Fajardo Perez M, Perez Herrero M. Serratus-intercostal interfascial plane block: alternative analgesia for open nephrectomy? Minerva Anestesiol. 2018 Jul;84(7):872-873. doi: 10.23736/S0375-9393.18.12808-2. Epub 2018 Feb 22. No abstract available. PMID 29479932
- [Background] Fernandez Martin MT, Lopez Alvarez S, Perez Herrero MA. Serratus-intercostal interfascial block as an opioid-saving strategy in supra-umbilical open surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Oct;65(8):456-460. doi: 10.1016/j.redar.2018.03.007. Epub 2018 May 20. English, Spanish. PMID 29789137